CLINICAL TRIAL: NCT07149727
Title: The Effect of Immersive Game Experience on Preoperative Anxiety and Compliance in Children Undergoing Supernumerary Tooth Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: YiHong Shao (Other)
Responsible Party: Sponsor-Investigator, YiHong Shao, Resident Physician, Department of Head and Neck Surgery,, Affiliated Hospital of Jiaxing University
Organization: Affiliated Hospital of Jiaxing University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-LP-004
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Supernumerary Teeth
Keywords: Teeth; Preoperative Anxiety; Pediatric Dentistry; Immersive Game; Behavioral Intervention
MeSH Terms: conditions — Tooth, Supernumerary | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): Participants receive standard preoperative care, including environmental temperature control, preoperative psychological counseling, and parent-guided distraction.
  Interventions: Other: Standard Care
- Intervention Group (Active Comparator): Participants receive standard care plus immersive game experience.
  Interventions: Behavioral: Immersive Game Experience (IGE)

INTERVENTIONS:
Other: Standard Care — Environmental temperature control, preoperative psychological counseling, and parent-guided distraction.
  Arms: Control Group
Behavioral: Immersive Game Experience (IGE) — Standard care plus immersive game experience, including role-playing scenarios (e.g., using dolls to simulate IV puncture), parent-child interactive games, environmental adjustments (children's music, colorful objects), and post-intervention rewards (cartoon stickers).
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to evaluate whether immersive game experience (IGE) can improve preoperative anxiety, compliance, and parental satisfaction in children aged 4-12 years undergoing supernumerary tooth extraction under general anesthesia. The main questions are:

Does IGE reduce anxiety measured by SCARED scores, heart rate, salivary cortisol, and LF/HF ratio?

Does IGE improve children's compliance and parental satisfaction?

Participants are randomized 1:1 to standard care or standard care plus IGE, which includes role-playing, parent-child interactive games, environmental adjustments, and rewards. Written informed consent is obtained from legal guardians, and all procedures follow ethical guidelines approved by Jiaxing First Hospital Ethics Committee (2025-LP-044). Outcomes are assessed by blinded staff using validated scales and physiological measures.

DETAILED DESCRIPTION:
The goal of this clinical trial is to evaluate whether immersive game experience (IGE) can improve preoperative emotional management, compliance, and parental satisfaction in children undergoing supernumerary tooth extraction. The main questions it aims to answer are:

Does immersive game experience reduce preoperative anxiety as measured by SCARED scores, heart rate, salivary cortisol, and LF/HF ratio?

Does immersive game experience improve children's compliance (Frankl compliance score) and parental satisfaction?

If there is a comparison group: Researchers will compare the control group receiving standard care (including environmental temperature control, preoperative psychological counseling, and parent-guided distraction) with the intervention group receiving standard care plus immersive game experience, to see if the intervention improves anxiety management, compliance, and satisfaction.

Participants will:

Be children aged 4-12 years undergoing supernumerary tooth extraction under general anesthesia, diagnosed by panoramic X-ray and/or CBCT;

Meet inclusion criteria: ASA physical status I or II, no sensory impairments, no diagnosed psychiatric or neurodevelopmental disorders, legal guardians able to provide informed consent, and children able to understand basic instructions;

Be excluded if they require emergency surgery, have significant developmental delays or cognitive impairment, history of severe sedation/anesthesia adverse events, active systemic infection or fever (>38°C) at admission, legal guardians with cognitive impairment or unable to complete questionnaires, or children refuse participation after initial explanation;

Be randomized 1:1 into control (n=52) or intervention group (n=50) using a computer-generated random number table with allocation concealment by opaque sealed envelopes; randomization performed by an independent researcher.

Interventions:

Control group: Standard care including environmental adjustments, psychological preparation, and parental guidance for distraction.

Intervention group: Standard care plus immersive game experience (IGE) including role-playing scenarios (e.g., using dolls to simulate IV puncture), parent-child interactive games (role reversal exercises), environmental adjustments (children's music, colorful objects), and rewards (cartoon stickers) after intervention.

Protection of human subjects:

Written informed consent obtained from legal guardians; child patient data kept confidential; gender-sensitive procedures conducted with guardian or same-gender staff present; independent in-hospital complaint channel established; staff trained regularly in minors' rights and emergency handling.

Statistical analysis:

IBM SPSS 22.0 and R 4.3.1 were used. Sample size calculation based on pretest SCARED score differences (power 90%, α=0.05, two-sided) yielded 102 participants considering 10% dropout. Continuous variables expressed as mean ± SD; categorical variables as frequency (percentage). Baseline comparisons by independent t-test or chi-square test. Primary outcomes (heart rate, SCARED scores, cortisol, LF/HF ratio) analyzed using repeated-measures ANOVA; secondary outcomes (Frankl compliance, satisfaction) analyzed using Mann-Whitney U, t-test, or chi-square test. Correlations by Pearson coefficient; multiple comparisons adjusted by Benjamini-Hochberg FDR. Moderator effects analyzed with group × SCARED interaction, adjusting for age and baseline anxiety. Significance defined as P<0.05.

Other specifications:

Approved by Jiaxing First Hospital Ethics Committee (2025-LP-044) and follows CONSORT guidelines.

All game props disinfected after use; physiological data collected after 5-min rest; saliva stored at -80°C and analyzed by high-sensitivity ELISA; compliance assessed by blinded surgeons. The study is monitored by the ethics committee, and major protocol changes require re-approval.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with impacted supernumerary teeth by panoramic radiograph and/or cone-beam CT (CBCT)
* ASA physical status I or II
* No sensory, auditory, or visual impairments
* No diagnosed psychiatric or neurodevelopmental disorders
* Legal guardian able to understand the study and provide written informed consent
* Child able to understand basic instructions

Exclusion Criteria:

* Require emergency surgery
* Significant developmental delay or cognitive impairment
* History of severe adverse reaction to sedation/anesthesia
* Active systemic infection or fever (>38°C) at admission
* Legal guardian with cognitive impairment or unable to complete questionnaires
* Child refuses participation after explanation

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Screen for Child Anxiety Related Emotional Disorders (SCARED) | Before intervention and preoperative period
  Anxiety level of children will be assessed using the Screen for Child Anxiety Related Emotional Disorders (SCARED) questionnaire, which contains 41 items scored on a 3-point Likert scale (0 = Not True or Hardly Ever True, 1 = Somewhat True or Sometimes True, 2 = Very True or Often True). The total score ranges from 0 to 82, with higher scores indicating greater anxiety severity (worse outcome).
Heart Rate | Before intervention and preoperative period
  Heart rate monitored to assess physiological anxiety response during the preoperative period.
Salivary Cortisol | Before intervention and preoperative period
  Cortisol concentration measured using high-sensitivity ELISA to evaluate stress response.

SECONDARY OUTCOMES:
Frankl Compliance Rating | During preoperative intervention and procedure
  Children's compliance during preoperative procedures rated using the Frankl Behavioral Rating Scale.
Parental Satisfaction | Immediately after procedure
  Parents' satisfaction with the preoperative intervention assessed using a standardized questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiaxing University Affiliated Hospital, Jiaxing, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No